CLINICAL TRIAL: NCT00195793
Title: A Multicenter, Randomized, Double-Blind, Prospective, Parallel Study to Compare the Safety and Efficacy of Fenofibrate or Ezetimibe as Add-On Therapy to Atorvastatin in Subjects With Combined Hyperlipidemia, Typical of the Metabolic Syndrome
Brief Title: A 16 Week Comparative Study of Fenofibrate Versus Ezetimibe as Add-on Therapy to Atorvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-661
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; fenofibrate; ezetimibe; atorvastatin
MeSH Terms: conditions — Hyperlipidemias | interventions — Fenofibrate; Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fenofibrate
Drug: ezetimibe
Drug: atorvastatin

SUMMARY:
The objective of this study is to evaluate the effects of adding Tricor 145 mg to once daily atorvastatin 20 mg on CHD lipid laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >= 18 years of age, any race, and any gender.
* Subjects must have the following fasting parameters:

  * LDL-C > 100 mg/dL and < 190 mg/dL.
  * TG level >= 175 mg/dL and < 1000 mg/dL.
  * HDL-C < 40 mg/dL (men) and < 50 mg/dL (women).
* Subjects must have one or more of the following:

  * Treated or untreated hypertension defined as blood pressure (BP)
  * 130 mmHg >= 85 mmHg (systolic / diastolic).
  * Waist circumference > 88 cm (35 inches) for women or > 102 cm (40 inches) for men.
  * Fasting glucose defined as >= 100 mg/dL but <= 125 mg/dL.
* Subject has, in the opinion of the investigator, a life expectancy greater than 6 months.
* Female subjects must have a negative pregnancy test prior to study enrollment.
* Female subjects of child bearing potential must agree to practice an effective barrier method of birth control for the duration of the study.
* Subject must be willing to observe the Step I Diet recommended by the NCEP throughout the study.
* Subject must be willing to participate in the study and to complete all follow-up assessments.

Exclusion Criteria:

* Subject has a known hypersensitivity to fenofibrate, ezetimibe, or atorvastatin
* Subject has been previously enrolled in this study.
* Subject has used an investigational drug within 30 days of study entry.
* Subject has been diagnosed with Type I or Type II Diabetes Mellitus or is currently being treated with anti-diabetic medication, or has a fasting glucose >= 126 mg/dL.
* Subject has a history of pancreatitis or cholelithiasis or a history of gastric or duodenal ulcer within 3 months of study entry.
* Subject has hematologic, digestive, or central nervous system disorder including cerebrovascular disease or degenerative disease that would limit study evaluation or participation.
* Subject has had a myocardial infarction, coronary bypass surgery, or angioplasty within 6 months of study entry.
* Subject has unstable or severe peripheral artery disease within 3 months of study entry.
* Subject has unstable angina pectoris or uncontrolled cardiac arrhythmias.
* Subject has congestive heart failure (CHF) as defined by NYHA Class III or IV
* Subject has coagulopathy (PT or PTT > 1.25 times control).
* Subject has known impairment of renal function (serum creatinine > 1.5 mg/dL), dysproteinemia, nephrotic-range proteinuria, or other renal disease.
* Subject has active or chronic hepatobiliary or hepatic disease (subjects with AST or ALT > 2 times the upper limit of the central laboratory reference range).
* Subject is pregnant or lactating.
* Subject is receiving hormonal therapy.
* Subject has a known history of thyroid disease or other endocrine abnormality.
* Subject has a history of diagnosed hereditary or acquired myopathy.
* Subject is known to be HIV positive.
* Subject has a history of mental instability, drug or alcohol (as defined by greater than 14 drinks per week) abuse, or subject has been treated for severe psychiatric illness, which, in the opinion of the investigator, may interfere with optimal participation in the study.
* Subject has received a solid organ transplant.
* Subject has a clinically significant, unstable, uncontrolled disease that could be adversely affected by study participation.
* Subject is unwilling or unable to consent to enter the study.
* Subject is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Percent change from Combination Baseline to 12 weeks post-Combination Baseline in direct measured HDL-C and TG. | Week 12

SECONDARY OUTCOMES:
Advanced lipid and inflammatory parameters | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott